CLINICAL TRIAL: NCT01236040
Title: Immunogenicity and Safety Study of GSK Biologicals' Cell Culture Derived Pandemic Influenza Vaccines GSK2590066A and GSK2592984A Administered to Healthy Adults 18 - 49 Years Old
Brief Title: Immunogenicity and Safety of Pandemic Influenza Vaccines in Adults Aged 18 - 49 Years Old
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 114371
Record Dates: First submitted 2010-10-28; First posted 2010-11-08 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: H5N1; Influenza; Pandemic
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (6):
- Group A (Experimental): Subjects will receive 2 doses of a formulation of GSK2590066A vaccine at a 21-day interval.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2590066A
- Group B (Experimental): Subjects will receive 2 doses of a formulation of GSK2592984A vaccine at a 21-day interval.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2592984A
- Group C (Placebo Comparator): Subjects will receive 2 doses of a placebo at a 21-day interval.
  Interventions: Other: Placebo
- Group D (Experimental): Subjects will receive 2 doses of a formulation of GSK2590066A vaccine at a 21-day interval.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2590066A
- Group E (Experimental): Subjects will receive 2 doses of a formulation of GSK2340274A vaccine at a 21-day interval.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2340274A
- Group F (Experimental): Subjects will receive 2 doses of a formulation of GSK2340273A vaccine at a 21-day interval.
  Interventions: Biological: GSK Biologicals' investigational vaccine GSK2340273A

INTERVENTIONS:
Biological: GSK Biologicals' investigational vaccine GSK2590066A — Intramuscular injection, two doses
  Arms: Group A; Group D
Biological: GSK Biologicals' investigational vaccine GSK2592984A — Intramuscular injection, two doses
  Arms: Group B
Biological: GSK Biologicals' investigational vaccine GSK2340274A — Intramuscular injection, two doses
  Arms: Group E
Biological: GSK Biologicals' investigational vaccine GSK2340273A — Intramuscular injection, two doses
  Arms: Group F
Other: Placebo — Intramuscular injection, two doses
  Other Names: Control
  Arms: Group C

SUMMARY:
This study will assess safety and immunogenicity of GSK Biologicals' H5N1 flu candidate vaccines GSK2590066A and GSK2340273A in healthy adults 18 - 49 years old.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject.
* Male and female adults, 18-49 years of age at the time of the first vaccination.
* Satisfactory baseline medical assessment by history and physical examination.
* Safety laboratory test results within the parameters specified in the protocol.
* Access to a consistent means of telephone contact
* Female subjects of non-childbearing potential may be enrolled in the study. Female subjects of childbearing potential may be enrolled in the study, if the subject: has practiced adequate contraception for 30 days prior to vaccination, and has a negative urine pregnancy test on the day of first vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Medical history of physician-confirmed infection with an H5N1 virus.
* Increased risk of occupational exposure to H5N1 influenza viruses.
* Previous vaccination at any time with an H5N1 vaccine, or with an oil-in water adjuvanted influenza vaccine.
* Planned administration of an adjuvanted influenza vaccine or an H5N1 pandemic vaccine during the entire study period.
* Use of any investigational or non-registered product other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness.
* Presence of neurological or psychiatric diagnoses which, although stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Evidence of current substance abuse, including alcohol, by medical history.
* Presence of a temperature >= 38.0ºC (≥100.4ºF), or acute symptoms greater than "mild" severity on the scheduled date of first dose.
* Diagnosed with cancer, or treatment for cancer, within 3 years. Persons with a history of cancer who are disease-free without treatment for 3 years or more are eligible.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Receipt of systemic glucocorticoids within 1 month prior to study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment.
* Receipt of any immunoglobulins and/or any blood products within 3 months of study enrollment or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin, outside of 24 hours prior to dosing, are eligible. Persons receiving prophylactic antiplatelet medications.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome.
* Administration of an inactivated seasonal influenza vaccine within 14 days before the first study vaccine dose, or of any other vaccine(s) not foreseen by the study protocol within 30 days before the first study vaccine dose. The administration of live attenuated trivalent seasonal influenza virus vaccine (LAIV) is allowed.
* Planned administration of any vaccine(s) not foreseen by the study protocol through completion of the Day 42 visit. The administration of LAIV is allowed.
* Any known or suspected allergy to any constituent of influenza vaccines or to latex, or history of severe reaction to a previous influenza vaccination.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin (β-hCG) test result prior to the first study vaccine dose.
* Lactating or nursing women.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 521 (Actual)
Dates: Start 2010-11-29 (Actual); Primary Completion 2011-09-06 (Actual); Study Completion 2012-08-20 (Actual)

PRIMARY OUTCOMES:
Immunogenicity with respect to components of the investigational vaccine Day 0 | Day 0
Immunogenicity with respect to components of the investigational vaccine Day 42 | Day 42
Occurrence of Grade 3 injection site pain | During a 7-day follow-up period (Day 0 to 6) after any vaccination

SECONDARY OUTCOMES:
Occurrence of each solicited local symptom | During a 7-day follow-up period (Day 0 to 6) after any vaccination
Occurrence of each solicited general symptom | During a 7-day follow-up period (Day 0 to 6) after any vaccination
Occurrence of unsolicited adverse events (AEs) | Within 21 days (Day 0 to 20) after any vaccination
Occurrence of AEs with medically attended visits (MAEs) | During the entire study period (from Day 0 to Month 12)
Occurrence and relationship to vaccination of (potential) immune mediated diseases (pIMDs) | During the entire study period (from Day 0 to Month 12)
Occurrence and relationship to vaccination of serious adverse events (SAEs) | During the entire study period (from Screening to Month 12)
Occurrence of adverse pregnancy outcomes | During the entire study period (from Day 0 to Month 12)
Clinical safety laboratory abnormalities | At Days 7, 28 and at Month 6.
Immunogenicity with respect to components of the investigational vaccine in terms of hemagglutinin Inhibition (HI) antibodies | At Days 0, 21, and 42 and Months 6 and 12
Immunogenicity with respect to components of the investigational vaccine in terms of microneutralization (MN) antibodies | Days 0, 21, and 42 and Months 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- United States (4):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Schuind A, Segall N, Drame M, Innis BL. Immunogenicity and Safety of an EB66 Cell-Culture-Derived Influenza A/Indonesia/5/2005(H5N1) AS03-Adjuvanted Vaccine: A Phase 1 Randomized Trial. J Infect Dis. 2015 Aug 15;212(4):531-41. doi: 10.1093/infdis/jiv091. Epub 2015 Feb 25. PMID 25722291
- See also: Results for study 114371 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/114371?search=study&#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 114371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114371 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register